CLINICAL TRIAL: NCT00323557
Title: Immuno-Augmentation With GM-CSF in Patients Receiving Pneumococcal Vaccine While Undergoing Treatment for Advanced Chronic Lymphocytic Leukemia (CLL)
Brief Title: Immuno-Augmentation With GM-CSF of Pneumococcal Vaccine in Chronic Lymphocytic Leukemia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0605
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Leukemia
Keywords: Chronic Lymphocytic Leukemia; Leukemia; Sargramostim; Pneumococcal Pneumonia; Pneumococcal Vaccine; Prevnar; GM-CSF; CLL
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Pneumonia, Pneumococcal | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pneumococcal Vaccine + GM-CSF (Experimental): Vaccine subcutaneously + GM-CSF (3 Doses of 250 mg subcutaneously) given either Pre Vaccine at Day -7, Day -1 and Day 0 (day of pneumococcal vaccine) or Post Vaccine given at Day 0, Day +3 and Day +7.
  Interventions: Drug: Sargramostim (GM-CSF)
- Pneumococcal Vaccine Alone (Experimental): First vaccine dose subcutaneously, Day 0.
  Interventions: Biological: Pneumococcal Vaccine

INTERVENTIONS:
Drug: Sargramostim (GM-CSF) — Starting with 3 doses of 250 micrograms subcutaneously, either pre or post vaccine. For pre vaccine, GM-CSF on days -7 (+ 1 day) and -3 (+ 1 day), in the week prior to vaccination for pre-vaccination immune priming; 3rd dose on the day of vaccination (day 0); and for post-vaccine GM-CSF given simultaneously on day of vaccination (day 0) and 2 more doses Day +3 and Day +7 after pneumococcal vaccine.
  Other Names: Leukine; GM-CSF; Granulocyte macrophage colony stimulating factor -
  Arms: Pneumococcal Vaccine + GM-CSF
Biological: Pneumococcal Vaccine — Subcutaneously on Day 0
  Other Names: Prevnar
  Arms: Pneumococcal Vaccine Alone

SUMMARY:
The goal of this clinical research study is to see if Leukine(R) (sargramostim) improves the effectiveness of the pneumococcal vaccine, a medicine used to prevent pneumococcal pneumonia, in patients with chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
Sargramostim (also commonly called granulocyte macrophage colony stimulating factor - GM-CSF) is a medication used to stimulate the bone marrow production of white blood cells before a stem cell transplant, after chemotherapy or after a bone marrow transplant. Pneumococcal vaccine is a medication used to prevent infections caused by a bacteria called Streptococcus pneumoniae.

If you have not had a gammaglobulins test (a test to measure immunity against certain infectious diseases) measured within three months before the study begins, then this blood test will be done before you receive any study medications.

Women who are able to have children must have a negative urine pregnancy test before starting treatment.

After consenting to this study, you will be randomly assigned (as in the toss of a coin) to receive treatment with sargramostim in addition to the pneumococcal vaccine or to receive pneumococcal vaccine alone (Prevnar).

* If you are randomized to vaccine plus sargramostim group, you will receive an injection of sargramostim at the same time you receive the pneumococcal vaccine.
* If you are randomized to the vaccine alone group, you will receive the pneumococcal vaccine on the first day.

Blood tests will be performed on the day of the pneumococcal vaccination, and 4 weeks, 12 weeks and 24 weeks after vaccination. Each of the blood tests will require about 4 teaspoons of blood. These blood tests will measure your immunity to pneumococcal infection.

If after 6 months of your first vaccination your body is not able to show immunity to pneumococcal infection, you will receive a second dose either pneumococcal vaccine plus sargramostim or pneumococcal vaccine alone. Your immunity will be checked again at 4 weeks, 12 weeks, and 24 weeks after this second dose. Only 4 teaspoon of blood will be required for the tests.

You may be removed from the study if you have a severe allergic reaction to the sargramostim and/or pneumococcal vaccine. The total maximum time you will be on this is study is 24 months.

This is an investigational study. Both of the medications used in this study are approved by the FDA. Up to 50 patients may be treated on this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1) Patients in complete / partial remission or those with active Chronic lymphocytic leukemia (CLL) with Rai stage 0 to 4.

Exclusion Criteria:

1. Patients will not be entered while neutropenic (PMNs < 500 cells/mm3) or having received Rituximab within 6 months.
2. Patients will not be entered while febrile (Temperature > 38 degrees C) within 1 week.
3. Active infection.
4. Patients with known Human immunodeficiency virus (HIV) infection.
5. Known history of allergy to Granulocyte/ macrophage colony stimulating factor (GM-CSF) or pneumococcal vaccine.
6. Chemotherapy other than Campath, fludarabine, cyclophosphamide, in 4 weeks.
7. Patients who have previously received pneumococcal vaccine within the preceding 12 months.
8. Absolute lymphocyte count less than 500 cells/mm3.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Safdar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Safdar A, Rodriguez GH, Rueda AM, Wierda WG, Ferrajoli A, Musher DM, O'Brien S, Koller CA, Bodey GP, Keating MJ. Multiple-dose granulocyte-macrophage-colony-stimulating factor plus 23-valent polysaccharide pneumococcal vaccine in patients with chronic lymphocytic leukemia: a prospective, randomized trial of safety and immunogenicity. Cancer. 2008 Jul 15;113(2):383-7. doi: 10.1002/cncr.23561. PMID 18470901
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 9, 2004 to July 16, 2009. All participants were recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 39 enrolled participants, four (4) participants withdrew consent and three (3) were ineligible thus all seven (7) were excluded from the trial before assignment to Pneumococcal Vaccine and Granulocyte Macrophage Colony-Stimulating Factor (GM-CSF) related treatment groups.
Period: Overall Study
Arm/Group | Pneumococcal Vaccine + GM-CSF | Pneumococcal Vaccine Alone
Started | 25 (GM-CSF pre and post vaccine.) | 7
Completed | 24 | 7
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumococcal Vaccine + GM-CSF | Pneumococcal Vaccine Alone | Total
Number analyzed (Participants) | 25 | 7 | 32
Age Continuous [Median (Full Range); unit: years] | 70 [51 to 91] | 61 [57 to 77] | 68 (10) [51 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 13 | 4 | 17
Region of Enrollment [Number; unit: participants]
  United States | 25 | 7 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (With Increase) Immune Response to GM-CSF With a Pneumococcal Vaccine
Description: Response defined as 2-fold rise in anticapsular immunoglobulin G (IgG) when prevaccination titer is compared with levels post vaccination and with a final level of >0.5 ug/mL. Anti-pneumococcal immunoglobulin titers measured at baseline and 1 month after vaccine. Response determined by measuring serum IgG to capsular polysaccharides from 6 of the most common infecting serotypes of Streptococcus pneumoniae.
Time Frame: Baseline and at 1 month after vaccine.
Measure: Number; unit: participants
Groups:
- Pneumococcal Vaccine + Pre Vaccine GM-CSF: Vaccine subcutaneously + GM-CSF 3 Doses of 250 mg subcutaneously given pre vaccination Day -7, Day -1 and Day 0 (day of pneumococcal vaccine).
- Pneumococcal Vaccine + Post Vaccine GM-CSF: Vaccine subcutaneously + GM-CSF 3 Doses of 250 mg subcutaneously given Day 0 (day of pneumococcal vaccine), and post vaccination at Day +3 and Day +7.
- Pneumococcal Vaccine Alone: First vaccine dose subcutaneously, Day 0. No CM-CSF.
Arm/Group | Pneumococcal Vaccine + Pre Vaccine GM-CSF | Pneumococcal Vaccine + Post Vaccine GM-CSF | Pneumococcal Vaccine Alone
Number analyzed (Participants) | 13 | 12 | 7
participants
  Pneumococcal Serotype 4 | 0 (5) | 0 | 1
  Pneumococcal Serotype 6B | 1 | 1 | 0
  Pneumococcal Serotype 9V | 1 | 1 | 1
  Pneumococcal Serotype 14 | 2 (66) | 2 | 0
  Pneumococcal Serotype 19F | 2 | 0 | 1
  Pneumococcal Serotype 23F | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: 6 years and 6 months
Arm/Group | Pneumococcal Vaccine + GM-CSF | Pneumococcal Vaccine Alone
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/7
Other Adverse Events (participants affected / at risk) | 9/25 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pneumococcal Vaccine + GM-CSF (N=25) | Pneumococcal Vaccine Alone (N=7)
Pain and redness at injection site (Skin and subcutaneous tissue disorders) | 6 | 1
Palmar Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Low grade fever (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No